CLINICAL TRIAL: NCT01770431
Title: A Multicenter, Randomized, Paralleled Control Clinical Study Investigating Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma After Radical Hepatectomy
Brief Title: Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma After Radical Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE-201101
Record Dates: First submitted 2013-01-01; First posted 2013-01-17 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-03

CONDITIONS: Hepatic Carcinoma
Keywords: Huaier Granule;; After radical hepatectomy;; Prevention of Recurrence and Metastasis;; Safety.
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — huaier

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huaier Granule group (Experimental): Huaier Granule group; specifications: 20g / bag; manufacturer: Qidong Gaitianli Medicines Co., Ltd..
  Administration: the Huaier Granule Electuary should be orally taken from the 15th day after surgery. Usage: Huaier Granule Electuary is continuously taken three times per day, 20g per time, until 96 weeks after surgery or until study termination. The subjects should not take any other anticancer drugs or immunomodulatory agents, except for Huaier Granule.
  Interventions: Drug: Huaier Granule
- Bank-control group (No Intervention): Blank-control group, not taking Huaier Granule, other anticancer drugs, or immunomodulatory agents.
  During the study, patients who need antiviral therapy, in both the test group and control group, can be treated according to the therapeutic principles.

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granule is a traditional Chinese medicine, 20g / time, 3 times/day,Po.
  Other Names: Huaier
  Arms: Huaier Granule group

SUMMARY:
To evaluate the efficacy and safety of Huaier Granule for prevention of recurrence and metastasis of hepatocarcinoma after radical hepatectomy.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Paralleled control Clinical Study Investigating Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma after Radical Hepatectomy,to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 and ≤ 75 years, both male and female;
* Radical hepatectomy has been performed for hepatocellular carcinoma;
* The hepatocellular carcinoma has been confirmed by pathological examination;
* Barcelona clinic liver cancer(BCLC) stage A or B;
* Not receiving any preoperative anticancer drug;
* The liver and kidney function satisfies the following conditions within 15 days after surgery (excluding day 15): aspartate aminotransferase(AST), glutamic-oxalacetic transaminase(ALT)<3 upper limit of normal(ULN), total bilirubin≤2ULN, serum creatinine <1.5 ULN;
* Other laboratory tests meet the following requirements within 15 days after surgery (excluding day 15): Hb≥9g/dl, platelet count≥60×109/L, absolute neutrophil count>1.0×109/L;
* The expected survival time ≥ 12 weeks;
* The subjects volunteer to sign the informed consent.

Exclusion Criteria:

* Hepatocellular carcinoma patients who received non-radical hepatectomy;
* Non-hepatocellular carcinoma patients;
* Those with Child-Pugh C;
* Pregnant or lactating women;
* Those with active bleeding due to various reasons;
* Those with HIV infection or AIDS-associated diseases;
* Those with severe acute and chronic diseases;
* Those with severe diabetes;
* Those with serious infectious diseases;
* Those who can not take drugs by oral route;
* Drug abusers or those with psychological or mental diseases that may interfere with study compliance;
* Conditions that are considered not suitable for this study investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2011-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Professor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Q, Shu C, Laurence AD, Chen Y, Peng BG, Zhen ZJ, Cai JQ, Ding YT, Li LQ, Zhang YB, Zheng QC, Xu GL, Li B, Zhou WP, Cai SW, Wang XY, Wen H, Peng XY, Zhang XW, Dai CL, Bie P, Xing BC, Fu ZR, Liu LX, Mu Y, Zhang L, Zhang QS, Jiang B, Qian HX, Wang YJ, Liu JF, Qin XH, Li Q, Yin P, Zhang ZW, Chen XP. Effect of Huaier granule on recurrence after curative resection of HCC: a multicentre, randomised clinical trial. Gut. 2018 Nov;67(11):2006-2016. doi: 10.1136/gutjnl-2018-315983. Epub 2018 May 25. PMID 29802174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 39 hospitals in China between December 7, 2011 and December 31, 2014. 1044 patients met eligibility criteria and were randomly assigned at a 2:1 ratio: 696 in Huaier group and 348 patients in the blank control group.
Groups:
- Huaier Granule Group: Huaier Granule group; specifications: 20g / bag; manufacturer: Qidong Gaitianli Medicines Co., Ltd..
  Administration: the Huaier Granule Electuary should be orally taken from the 15th day after surgery. Usage: Huaier Granule Electuary is continuously taken three times per day, 20g per time, until 96 weeks after surgery or until study termination. The subjects should not take any other anticancer drugs or immunomodulatory agents, except for Huaier Granule.
  Huaier Granule: Huaier Granule is a traditional Chinese medicine, 20g / time, 3 times/day,Po.
- Bank-control Group: Blank-control group, not taking Huaier Granule, other anticancer drugs, or immunomodulatory agents.
  During the study, patients who need antiviral therapy, in both the test group and control group, can be treated according to the therapeutic principles.
  Huaier Granule: Huaier Granule is a traditional Chinese medicine, 20g / time, 3 times/day,Po.
Period: Overall Study
Arm/Group | Huaier Granule Group | Bank-control Group
Started | 696 | 348
Completed | 686 | 316
Not Completed | 10 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Huaier Granule Group | Bank-control Group | Total
Number analyzed (Participants) | 686 | 316 | 1002
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 573 | 275 | 848
  >=65 years | 113 | 41 | 154
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 61 | 182
  Male | 565 | 255 | 820
Region of Enrollment [Count of Participants; unit: Participants]
  China | 686 | 316 | 1002
Number of tumor [Count of Participants; unit: Participants]
  Single tumor | 595 | 274 | 869
  Multiple tumors | 91 | 42 | 133

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Recurrence and Metastasis After Hepatectomy
Description: At week 94 after took medicine, assess incidence of recurrence and metastasis after hepatectomy.
Time Frame: Week 94 after took medicine
Measure: Count of Participants; unit: Participants
Arm/Group | Huaier Granule Group | Bank-control Group
Number analyzed (Participants) | 686 | 316
Participants
  Recurrence-free | 428 | 155
  Recurrence | 258 | 161
Statistical Analysis 1: Comparison: Huaier Granule Group vs Bank-control Group; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; chi-squared = 14.7315

2. Secondary Outcome: Postoperative Survival Period
Description: Assess Postoperative survival period
Time Frame: Week 94 after took medicine
Measure: Median (Standard Error); unit: weeks
Arm/Group | Huaier Granule Group | Bank-control Group
Number analyzed (Participants) | 686 | 316
weeks | 75.5 (1.15) | 68.5 (1.89)
Statistical Analysis 1: Comparison: Huaier Granule Group vs Bank-control Group; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.55 to 0.81]

ADVERSE EVENTS:
Arm/Group | Huaier Granule Group | Bank-control Group
Serious Adverse Events (participants affected / at risk) | 0/686 | 0/316
Other Adverse Events (participants affected / at risk) | 35/686 | 6/316
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Huaier Granule Group (N=686) | Bank-control Group (N=316)
Diarrhea (Product Issues) | 35 (175) | 6 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days